CLINICAL TRIAL: NCT05775744
Title: Management of Postpartum Preeclampsia
Acronym: MOPP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Deepika Sagaram, MD, Assistant Clinical Professor, Rutgers, The State University of New Jersey
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro2022001222
Record Dates: First submitted 2023-02-17; First posted 2023-03-20 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-04

CONDITIONS: Postpartum Preeclampsia

STUDY DESIGN:
Intervention Model Description: The investigators will study and compare two cohorts of patients. The first is a retrospective cohort, including patients delivered at Robert Wood Johnson University Hospital and Cooperman Barnabas Medical Center. The second is a prospective cohort that will enroll patients immediately postpartum who are eligible for our treatment protocol.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prospective interventional arm (Experimental): The prospective cohort will identify patients in the postpartum period of their delivery hospitalization who are at risk of readmission for hypertensive disorders in the initial six weeks postpartum. Those at risk include patients with diagnosed with chronic hypertension or PIH. Chronic hypertension is defined as either taking antihypertensive medications or a blood pressure of greater than or equal to 140/90 mm Hg prior to 20 weeks of gestation. Pregnancy induced hypertension includes gestational hypertension, preeclampsia without severe features, preeclampsia with severe features and Hemolysis, Elevated Liver enzymes and Low Platelets (HELLP). The minimum requirement to be diagnosed with this spectrum of disorders is having two blood pressures of greater than or equal to 140/90 mm Hg during the antepartum, intrapartum or postpartum periods.
  Interventions: Other: Tight postpartum blood pressure control
- Retrospective observational arm (No Intervention): The retrospective cohort will include all patients diagnosed with chronic hypertension or pregnancy-induced hypertensive (PIH) disorders at Robert Wood Johnson University Hospital and Cooperman Barnabas Medical Center in the past two years, including those presenting to the Emergency Department or readmitted for hypertensive disorders, during the immediate six weeks postpartum.

INTERVENTIONS:
Other: Tight postpartum blood pressure control — The standard of care for patients with pregnancy induced hypertension is to start antihypertensive therapy if blood pressures are consistently over 150/100 mm Hg. There is no established standard of care for titrating blood pressure medication in the postpartum period for those with chronic hypertension and the approach to these patients varies by institution. The intervention in this study will be to start antihypertensive medications at a lower blood pressure cutoff, which is commonly used in the non-pregnant patient population to more tightly control blood pressure. Remote patient monitoring may be considered standard of care. The blood pressure targets chosen for this study are considered to be standard of care for non-pregnant people.
  Arms: Prospective interventional arm

SUMMARY:
The aim of this study is to assess the effect of a lower treatment threshold for antihypertensive medication and tighter blood pressure control, using remote blood pressure monitoring, on reducing Emergency Room visits for our postpartum patients with hypertensive disease.

DETAILED DESCRIPTION:
The aim of this study is to assess the effect of lower treatment threshold for initiating antihypertensive medication and tighter blood pressure control, using remote blood pressure monitoring, on reducing Emergency Room visits for our postpartum patients with hypertensive disease.

The investigators will study and compare two cohorts of patients. The first is a retrospective cohort, including patients delivered at Robert Wood Johnson University Hospital and Cooperman Barnabas Medical Center. The second is a prospective cohort that will enroll patients immediately postpartum who are eligible for our treatment protocol.

ELIGIBILITY:
Inclusion Criteria:

* Chronic hypertension, gestational hypertension, or preeclampsia.
* Delivery of a neonate after 20 weeks during their current hospitalization
* Able to consent
* 18 years old or above
* English or Spanish speaking
* Planning to follow up with a physician associated with Robert Wood Johnson University Hospital or Cooperman Barnabas Medical Center
* Ability to follow directions

Exclusion Criteria:

* Any medical condition that the providers feel is a contraindication to the MOPP algorithm.
* Planning to follow up with an outside institution.
* Unwillingness to take blood pressure at home.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 392 (Actual)
Dates: Start 2023-03-28 (Actual); Primary Completion 2024-03-26 (Actual); Study Completion 2024-03-26 (Actual)

PRIMARY OUTCOMES:
Postpartum Emergency Department visits for hypertensive disorders | Six weeks from date of delivery
  Any patient that returns to the Emergency Department for hypertensive disorders

SECONDARY OUTCOMES:
Postpartum readmissions for hypertensive disorders | 6 weeks form date of delivery
  Any patient that is readmitted to the hospital for hypertensive disorders.
Number of acute postpartum complications of preeclampsia | 6 weeks from date of delivery
  Postpartum complications include stroke, seizure, thrombocytopenia, elevated liver enzymes, liver rupture, kidney injury.
Lab abnormalities because of preeclampsia | 6 weeks from date of delivery
  Rate of lab abnormalities including acute kidney injury (creatinine >1.1 mg/dL), transaminitis (liver function tests > 2x upper limit of normal), or thrombocytopenia (platelet count < 100,000 uL)
Blood pressure at the postpartum visit | 6 weeks from date of delivery
  Measurement of blood pressure value at 6 week postpartum visit
Breastfeeding rates at 6 weeks postpartum | 6 weeks from date of delivery
  Rates of exclusive breastfeeding at 6 week postpartum visit.
Compliance with follow up at postpartum visits | 6 weeks from date of delivery
  If patient shows up to postpartum visit or not
Composite maternal cardiovascular and other morbidity | One year from delivery
  Death, any new heart failure, stroke or encephalopathy, myocardial ischemia or angina, pulmonary edema, ICU admission/ intubation, encephalopathy, or renal failure.
Short-term cardiovascular disease | One year from delivery
  The effect of aggressive postpartum preeclampsia on incidents of cardiovascular diseases, which include coronary heart disease (acute myocardial infarction, ischemic heart disease, hypertensive heart disease, and congestive heart failure), and stroke (ischemic and hemorrhagic strokes).
Socioeconomic factors | One year from delivery
  The impact of race/ethnicity and insurance status on primary and secondary outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Deepika Sagaram, MD, Principal Investigator — Rutgers, Robert Wood Johnson
Locations (2):
- United States (2):
  - Cooperman Barnabas Medical Center, Livingston, New Jersey
  - Robert Wood Johnson Medical School, New Brunswick, New Jersey

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data will be provided to those inquiries to the corresponding author of the manuscript if published. If no manuscript is published, inquiries can be directed to the principal investigator.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will be available on publication and will remain available for two years.
Access Criteria: The principal investigator will individually assess all requests for data.

REFERENCES:
- [Background] Patel S, Rodriguez AN, Macias DA, Morgan J, Kraus A, Spong CY. A Gap in Care? Postpartum Women Presenting to the Emergency Room and Getting Readmitted. Am J Perinatol. 2020 Dec;37(14):1385-1392. doi: 10.1055/s-0040-1712170. Epub 2020 May 30. PMID 32473598
- [Background] Bruce KH, Anderson M, Stark JD. Factors associated with postpartum readmission for hypertensive disorders of pregnancy. Am J Obstet Gynecol MFM. 2021 Sep;3(5):100397. doi: 10.1016/j.ajogmf.2021.100397. Epub 2021 May 12. PMID 33991709
- [Background] Podymow T, August P. Postpartum course of gestational hypertension and preeclampsia. Hypertens Pregnancy. 2010;29(3):294-300. doi: 10.3109/10641950902777747. PMID 20670153
- [Background] Fasanya HO, Hsiao CJ, Armstrong-Sylvester KR, Beal SG. A Critical Review on the Use of Race in Understanding Racial Disparities in Preeclampsia. J Appl Lab Med. 2021 Jan 12;6(1):247-256. doi: 10.1093/jalm/jfaa149. PMID 33227139
- [Background] Hypertension in pregnancy. Report of the American College of Obstetricians and Gynecologists' Task Force on Hypertension in Pregnancy. Obstet Gynecol. 2013 Nov;122(5):1122-1131. doi: 10.1097/01.AOG.0000437382.03963.88. No abstract available. PMID 24150027
- [Background] Whelton PK, Carey RM, Aronow WS, Casey DE Jr, Collins KJ, Dennison Himmelfarb C, DePalma SM, Gidding S, Jamerson KA, Jones DW, MacLaughlin EJ, Muntner P, Ovbiagele B, Smith SC Jr, Spencer CC, Stafford RS, Taler SJ, Thomas RJ, Williams KA Sr, Williamson JD, Wright JT Jr. 2017 ACC/AHA/AAPA/ABC/ACPM/AGS/APhA/ASH/ASPC/NMA/PCNA Guideline for the Prevention, Detection, Evaluation, and Management of High Blood Pressure in Adults: A Report of the American College of Cardiology/American Heart Association Task Force on Clinical Practice Guidelines. Hypertension. 2018 Jun;71(6):e13-e115. doi: 10.1161/HYP.0000000000000065. Epub 2017 Nov 13. No abstract available. PMID 29133356
- [Background] Tita AT, Szychowski JM, Boggess K, Dugoff L, Sibai B, Lawrence K, Hughes BL, Bell J, Aagaard K, Edwards RK, Gibson K, Haas DM, Plante L, Metz T, Casey B, Esplin S, Longo S, Hoffman M, Saade GR, Hoppe KK, Foroutan J, Tuuli M, Owens MY, Simhan HN, Frey H, Rosen T, Palatnik A, Baker S, August P, Reddy UM, Kinzler W, Su E, Krishna I, Nguyen N, Norton ME, Skupski D, El-Sayed YY, Ogunyemi D, Galis ZS, Harper L, Ambalavanan N, Geller NL, Oparil S, Cutter GR, Andrews WW; Chronic Hypertension and Pregnancy (CHAP) Trial Consortium. Treatment for Mild Chronic Hypertension during Pregnancy. N Engl J Med. 2022 May 12;386(19):1781-1792. doi: 10.1056/NEJMoa2201295. Epub 2022 Apr 2. PMID 35363951
- [Background] McManus RJ, Mant J, Haque MS, Bray EP, Bryan S, Greenfield SM, Jones MI, Jowett S, Little P, Penaloza C, Schwartz C, Shackleford H, Shovelton C, Varghese J, Williams B, Hobbs FD, Gooding T, Morrey I, Fisher C, Buckley D. Effect of self-monitoring and medication self-titration on systolic blood pressure in hypertensive patients at high risk of cardiovascular disease: the TASMIN-SR randomized clinical trial. JAMA. 2014 Aug 27;312(8):799-808. doi: 10.1001/jama.2014.10057. PMID 25157723
- [Background] Chen TY, Kao CW, Cheng SM, Chang YC. Effect of Home Medication Titration on Blood Pressure Control in Patients With Hypertension: A Meta-Analysis of Randomized Controlled Trials. Med Care. 2019 Mar;57(3):230-236. doi: 10.1097/MLR.0000000000001064. PMID 30762831
- [Background] Hirshberg A, Sammel MD, Srinivas SK. Text message remote monitoring reduced racial disparities in postpartum blood pressure ascertainment. Am J Obstet Gynecol. 2019 Sep;221(3):283-285. doi: 10.1016/j.ajog.2019.05.011. Epub 2019 May 20. No abstract available. PMID 31121137
- [Background] Hoppe KK, Williams M, Thomas N, Zella JB, Drewry A, Kim K, Havighurst T, Johnson HM. Telehealth with remote blood pressure monitoring for postpartum hypertension: A prospective single-cohort feasibility study. Pregnancy Hypertens. 2019 Jan;15:171-176. doi: 10.1016/j.preghy.2018.12.007. Epub 2018 Dec 31. PMID 30825917
- [Background] Austin PC. An Introduction to Propensity Score Methods for Reducing the Effects of Confounding in Observational Studies. Multivariate Behav Res. 2011 May;46(3):399-424. doi: 10.1080/00273171.2011.568786. Epub 2011 Jun 8. PMID 21818162
- [Background] Lash TL, Fox MP, MacLehose RF, Maldonado G, McCandless LC, Greenland S. Good practices for quantitative bias analysis. Int J Epidemiol. 2014 Dec;43(6):1969-85. doi: 10.1093/ije/dyu149. Epub 2014 Jul 30. PMID 25080530